CLINICAL TRIAL: NCT00954330
Title: Surgical Versus Functional Treatment for Acute Ruptures of the Lateral Ligament Complex of the Ankle in Young Males - A Randomized Controlled Trial With a Mean of 14 Years Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Defense Forces (Other Government)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 555555
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Ankle Injury
Keywords: rct, intervention, surgery, lateral ligament injury of the ankle; REturn to pre-injury level
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery (Experimental): All twenty-five patients underwent ligament repair, where the ruptured ends of the FTA (in 11 cases) or FTA and FC (in 14 cases) ligaments were rejoined by using absorbable sutures. A supine position and a tourniquet were used. A curvilinear skin incision of 5-10 cm was made; the retinacular structures were incised and the hematoma was removed.
  Interventions: Procedure: lateral ligament surgery
- functional treatment (Active Comparator): Twenty-six patients randomized to the functional treatment received a functional light-weight orthotic device (Air-Cast ankle brace, Summit, New Jersey) for 3 weeks. Full weight bearing was allowed. The ankle brace allowed dorsi- and plantarflexion but it restricted inversion and eversion of the ankle
  Interventions: Device: functional treatment

INTERVENTIONS:
Procedure: lateral ligament surgery — . The disrupted FTA or/and FC and superficial retinacular structures were repaired by using absorbable sutures. In case of avulsion from the bone, the ligament was reapproximated with the use of sutures that were passed through 2.0 millimeter drill-holes in the bone.
  Arms: surgery
Device: functional treatment — Twenty-six patients randomized to the functional treatment received a functional light-weight orthotic device (Air-Cast ankle brace, Summit, New Jersey) for 3 weeks. Full weight bearing was allowed. The ankle brace allowed dorsi- and plantarflexion but it restricted inversion and eversion of the ankle.
  Arms: functional treatment

SUMMARY:
The aim of this prospective randomized controlled trial was to compare the effectiveness of surgical and conservative treatment in acute lateral ligament injury of ankle. The more detailed aims were to assess the function, physical activity level, re-injuries, objective stability and radiographic changes seen by magnetic resonance imaging in patients randomized to surgery or to functional treatment after a mean of 14 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included positive stress radiographs (in all cases) and arthrography 15 (5 cases) proven fibulotalar anterior (FTA) and fibulocalcanear (FC) ligament injury.
* The positive findings for a lateral ligament injury included a clinically unstable ankle and a radiological talar tilt >6 degrees or ADS >5 mm compared with the uninjured opposite ankle.

Exclusion Criteria:

* The exclusion criteria for the study were diabetes, inflammatory arthritis, previous severe trauma, pre-existing instability of joints.
* In addition, patients were excluded from our study if they had previously undergone surgery of the ankle region.

Ages: 19 Years to 25 Years | Sex: Male
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 1991-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The main outcome measure in the present study was a validated ankle injury scoring scale, A Performance Test Protocol and Scoring Scale for the Evaluation of Ankle Injuries.

SECONDARY OUTCOMES:
Return to pre-injury level in physical activity, re-injuries of the same ankle, visits to physician due to the same ankle, range of joint motion, subjective satisfaction and complications were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Central military hospital, Helsinki, Finland